CLINICAL TRIAL: NCT01594047
Title: Perioperative Opioid-induced Hyperalgesia and Its Prevention With Ketamine and Methadone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Emiliano Tognoli, medical doctor, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: metadone
Record Dates: First submitted 2012-05-05; First posted 2012-05-08 (Estimated); Results first posted 2023-10-02 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Post Operative Pain; Hyperalgesia
Keywords: hyperalgesia; Patient controlled analgesia; morphine; methadone; ketamine
MeSH Terms: conditions — Pain, Postoperative; Hyperalgesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- zero/morphine (No Intervention): Patient received a standard balance anaesthesia and morphine for post operative pain.
- ketamine/morphine (Experimental): Ketamine infusion scheme: 5mcg/Kg/min from induction od anaesthesia for 10 min, than 2,5mcg/Kg/min for 20 min and than 2 mcg/Kg/min to the end of surgery.
  Interventions: Drug: ketamine infusion
- zero/metadone (Experimental): Methadone PCA
  Interventions: Drug: Methadone PCA
- ketamine/methadone (Experimental): Ketamine infusion scheme: 5mcg/Kg/min from induction od anaesthesia for 10 min, than 2,5mcg/Kg/min for 20 min and than 2 mcg/Kg/min to the end of surgery.
  Methadone administered by a PCA system (dose 2 mg, lock-out 12min.).
  Interventions: Drug: ketamine infusion; Drug: Methadone PCA

INTERVENTIONS:
Drug: ketamine infusion — Ketamine infusion scheme: 5mcg/Kg/min from induction od anaesthesia for 10 min, than 2,5mcg/Kg/min for 20 min and than 2 mcg/Kg/min to the end of surgery
  Other Names: hyperalgesia-blocker
  Arms: ketamine/methadone; ketamine/morphine
Drug: Methadone PCA — Methadone administered by a PCA system (dose 2 mg, lock-out 12min.)
  Other Names: hyperalgesia-blocker
  Arms: ketamine/methadone; zero/metadone

SUMMARY:
Background: In perioperative period inhibition of N-Methyl-D-Aspartate receptor prevents opioid-induced hyperalgesia and reduce postoperative opioid requirement after abdominal surgery. Methadone is both a µ-opioid receptor agonist like Morphine and a N-Methyl-D-Aspartate antagonist. Study Aim. To evaluate the efficacy of intraoperative Ketamine and postoperative Methadone analgesia in preventing opioid-induced hyperalgesia after abdominal surgery.

DETAILED DESCRIPTION:
not desired

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing open colo-rectal surgery

Exclusion Criteria:

* ASA status more than II, history of chronic pain, ischemic heart disease or chronic pulmonary disease, allergy to any drugs used in the protocol. Body Max Index more than 35.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2009-12-01 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2014-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Tognoli, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

REFERENCES:
- [Derived] Tognoli E, Proto PL, Motta G, Galeone C, Mariani L, Valenza F. Methadone for postoperative analgesia: contribution of N-methyl-D-aspartate receptor antagonism: A randomised controlled trial. Eur J Anaesthesiol. 2020 Oct;37(10):934-943. doi: 10.1097/EJA.0000000000001217. PMID 32516227

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine/Methadone: Ketamine infusion scheme: 5mcg/Kg/min from induction od anaesthesia for 10 min, than 2,5mcg/Kg/min for 20 min and than 2 mcg/Kg/min to the end of surgery.
  Methadone administered by a PCA system (dose 2 mg, lock-out 12min.).
  ketamine infusion: Ketamine infusion scheme: 5mcg/Kg/min from induction od anaesthesia for 10 min, than 2,5mcg/Kg/min for 20 min and than 2 mcg/Kg/min to the end of surgery
  Methadone PCA: Methadone administered by a PCA system (dose 2 mg, lock-out 12min.)
Period: Overall Study
Arm/Group | Zero/Morphine | Ketamine/Morphine | Zero/Metadone | Ketamine/Methadone
Started | 29 | 30 | 27 | 27
Completed | 24 | 25 | 23 | 24
Not Completed | 5 | 5 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zero/Morphine | Ketamine/Morphine | Zero/Metadone | Ketamine/Methadone | Total
Number analyzed (Participants) | 24 | 25 | 23 | 24 | 96
Age, Continuous [Mean (Full Range); unit: years] | 58 [40 to 75] | 60 [46 to 75] | 57 [42 to 70] | 57 [34 to 71] | 58 [34 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 8 | 10 | 33
  Male | 15 | 19 | 15 | 14 | 63

OUTCOME MEASURES:

1. Primary Outcome: the Extent of Hyperalgesia Area Proximal to Surgical Wound
Description: Hyperalgesia is determined by stimulating with a won Fray hair N°16 along three lines at a right angle to the top, middle, and bottom sides of the surgical incision. Each line starts from the edge of the abdomen to the surgical incision.
  Stimulation continue from the edge toward the surgical incision until the patients reported a worsening in sensation The distance from the incision to where sensation change was measured. The mean of the three assessments was used as a measure of the extent of the hyperalgesia area.
Time Frame: 24 and 48 hours after surgery
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Zero/Morphine | Ketamine/Morphine | Zero/Metadone | Ketamine/Methadone
Number analyzed (Participants) | 24 | 25 | 23 | 24
cm
  24 hours | 19.5 (12.76) | 14.68 (13.04) | 15.28 (12.72) | 11.04 (11.13)
  48 hours | 16.04 (13.23) | 16.38 (14.05) | 18.09 (15.34) | 14.51 (12.75)

2. Secondary Outcome: Pain Intensity Measured by a Numeric Rating Scale (NRS)
Description: A Numerical Rating Scale (NRS) from 0 to 10 is used as a measure of pain intensity. Zero indicates the absence of any pain and 10 the worse pain never felt.
Time Frame: 24 and 48 hours after surgery
Population: We performed a Dunn multiple comparison test for specific comparisons to assess group differences compared with the control group (0-Mo). Notably, the interaction term allowed us to test whether the effect of the two drugs, when jointly administered, was additive (lack of interaction) or more/ less than additive (presence of interaction). Data at 24 and 48 h were analyzed separately.
Measure: Mean (Standard Deviation); unit: units on NRS
Arm/Group | Zero/Morphine | Ketamine/Morphine | Zero/Metadone | Ketamine/Methadone
Number analyzed (Participants) | 24 | 25 | 23 | 24
units on NRS
  NRS static 24 hours | 1.92 (1.38) | 1.64 (1.32) | 0.61 (1.03) | 0.78 (1.28)
  NRS dynamic 24 hours | 4.75 (1.80) | 4.68 (1.95) | 3.13 (2.20) | 3.04 (1.66)
  NRS static 48 hours | 1.36 (1.92) | 0.88 (1.13) | 0.87 (1.36) | 0.5 (0.88)
  NRS dynamic 48 hours | 4.27 (1.86) | 4.44 (1.42) | 2.65 (1.92) | 2.75 (1.96)

3. Secondary Outcome: Opioid Consumption
Description: Cumulative opioid consumption at 48 hours from surgery ( end of the study)
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Zero/Morphine | Ketamine/Morphine | Zero/Metadone | Ketamine/Methadone
Number analyzed (Participants) | 24 | 25 | 23 | 24
mg | 56.09 (28.99) | 66.9 (29.37) | 43.64 (20.24) | 38.96 (20.95)

ADVERSE EVENTS:
Time Frame: For each patient, adverse event data were collected up to 48 hours from surgery ( end of the study)
Description: An adverse event is defined accordingly with the clinicaltrials.gov definitions.
Arm/Group | Zero/Morphine | Ketamine/Morphine | Zero/Metadone | Ketamine/Methadone
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
We chose to analyse mechanical static punctuate hyperalgesia along three lines lateral to the surgical wound, as it is the most common test used to characterise the effect of ketamine and others NMDAr blockers on neuroplasticity in surgical patients. We are aware that there is increasing evidence that the quantitative sensory testing may be more effective and specific in detecting and defining hyperalgesia, both in acute and chronic settings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes